CLINICAL TRIAL: NCT04112654
Title: Prospective Randomized Evaluation of the Contribution of Low-pressure Intra-abdominal Insufflation for Laparoscopic Colic Resection
Brief Title: Evaluation of the Contribution of Low-pressure Intra-abdominal Insufflation for Laparoscopic Colic Resection
Acronym: LoPreCol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOPRECOL-IPC 2017-02; LOPRECOL-IPC 2017-02 (Other: Sponsor)
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Colonic Disease
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional laparoscopy (Active Comparator): Laparoscopy realized at the conventional pressure (12-15 mmHg) using conventional insufflator.
  Interventions: Procedure: Conventional pressure laparoscopy
- Low pressure laparoscopy (Experimental): Laparoscopy realized at low pressure (6-8mmHg) using pressure-controlled insufflator AirSeal®
  Interventions: Procedure: Low pressure laparoscopy

INTERVENTIONS:
Procedure: Conventional pressure laparoscopy — Conventional pressure laparoscopy using conventional insufflator AirSeal®
  Arms: Conventional laparoscopy
Procedure: Low pressure laparoscopy — Low pressure laparoscopy using pressure-controlled insufflator AirSeal®
  Arms: Low pressure laparoscopy

SUMMARY:
The laparoscopic surgery requires gas insufflation in the peritoneal cavity and the operator chooses the intraabdominal insufflation pressure. In general, during a conventional laparoscopy, this pressure is 12 to 15 mmHg. The reduction of the intra-abdominal pressure minimizes the parietal trauma due to the insufflation and could lead to a reduction of the postoperative pains and could allow an earlier recovery. In this study, the investigator propose to evaluate the benefits of a low pressure insufflation (6-8 mmHg) with pressure-controlled insufflator in patients with a mild or malignant colon pathology requiring surgical colic resection. The main objective of the study is to demonstrate that the laparoscopic colic resection at low pressure reduces the theoretical hospital stay of one day compared to the conventional laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Colic lesion justifying surgical resection by segmental colectomy,
* Surgery proposed by laparoscopy,
* Body mass index (BMI) ≤30 kg/m2,
* Written informed consent signed by the patient,
* Patient affiliated to the national French statutory healthcare insurance, system or beneficiary of this regimen.

Exclusion Criteria:

* Probable realization of a stoma during the procedure,
* Robot-assisted approach,
* Contraindication to laparoscopic surgery,
* Pregnant or likely to be pregnant,
* Patient deprived of liberty or placed under the authority of a tutor,
* Patient considered geographically socially or psychologically unable to comply with the study procedure and the medical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
The theoretical hospital stay | from hospitalization day until hospital discharge, assessed up to 15 days
  The theoretical hospital stay in days (calculated from the day of the surgery to the theoretical day of discharge according to predefined exit criteria)

SECONDARY OUTCOMES:
Morbidity rate | 20 days post surgery
  Morbidity evaluated according Dindo-clavien classification
Mortality rate | 20 days post surgery
  Dead patient listing
GastroIntestinal-Quality-of-Life Index (GIQLI) | 20 days and 3 months post surgery
  GastroIntestinal-Quality-of-Life Index (GIQLI) questionnaire, 36 questions, each containing 4 answers equating to a score ranging from 0 (least desirable answer) to 4 (most desirable answer). Total score range 0-144.
Short Form Health (SF12) score | 20 days and 3 months post surgery
  This questionnaire is an abbreviated version of the "Medical Outcomes Study Short-Form General Health Survey" (SF-36) contains only 12 items out of 36 with minimum score 0 (bad quality life) and maximum score at 100 (good quality life).
Pain score using self-report pain assessment tool (EVA) | From surgery to hospital discharge assessed up to 15 days, at 20 days and at 3 months post surgery
  EVA measures the intensity of pain on a scale of 0 (no pain) to 10 (maximum pain imaginable)
Intestinal transit recovery time frame | From surgery to transit recovery assessed up to 15 days
  Period duration from surgery to intestinal gas recovery time (in days)
Nausea and vomiting incidence | From surgery to hospital discharge assessed up to 15 days
  Nausea and vomiting listing
Analgesic treatment incidence | From surgery to 3 months post surgery
  Non-morphine and morphine analgesic consumption
Real hospitalization duration | From hospitalization day until hospital discharge assessed up to 15 days
  Real hospitalization duration (actual patient discharge date based on non-medical criteria)
Rehospitalization number | from hospital discharge assessed up to 15 days to 3 months post surgery
  Rehospitalization listing
Differential cost of patient care | From surgery to hospital discharge assessed up to 15 days
  According operating room occupation and real hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Cecile DE CHAISEMARTIN, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France